CLINICAL TRIAL: NCT00616291
Title: Immunotherapy of Patients With Androgen-Independent Prostate Carcinoma Using NY-ESO-1/LAGE1 Peptide Vaccine (SPORE #: 11-01-30-14)
Brief Title: Vaccine Therapy in Treating Patients With Metastatic, Progressive Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Teresa Hayes, Associate Professor, Baylor College of Medicine
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000579579; P50CA058204 (NIH); BCM-H-17274; BCM-SPORE-11-01-30-14; NCT00711334 (obsolete NCT alias)
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (3):
- Group I (Experimental): MHC Class I binding peptide at 1000 mcg
  Interventions: Biological: NY-ESO-1/LAGE-1 HLA class I/II peptide vaccine
- Group II (Experimental): MHC Class II binding peptide at 1000 mcg
  Interventions: Biological: NY-ESO-1/LAGE-1 HLA class I/II peptide vaccine
- Group III (Experimental): Combination MHC Class I and II binding peptide at 1000 mcg each
  Interventions: Biological: NY-ESO-1/LAGE-1 HLA class I/II peptide vaccine

INTERVENTIONS:
Biological: NY-ESO-1/LAGE-1 HLA class I/II peptide vaccine

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects of a peptide vaccine in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and tolerance of NY-ESO-1/LAGE-1 class-I and class-II vaccine administered subcutaneously in patients with androgen-independent metastatic prostate cancer.

Secondary

* Compare the response induced by immunotherapy with a combined class-I and class-II NY-ESO-1/LAGE-1 vaccine to responses obtained to either class I or class II peptides alone.
* Evaluate whether the inclusion of class-II epitopes in a peptide vaccine will result in a better antitumor immune response than class-I epitopes alone.
* Determine antitumor activity by antigen response assays including cytokine elaboration, changes in frequency of peripheral T cells that recognize tumor, and intra/peritumoral cellular infiltrates and cytokine expression in responding and nonresponding metastasis.

OUTLINE: Patients receive NY-ESO-1/LAGE-1 peptide vaccine subcutaneously every other week for 12 weeks in the absence of disease progression or unacceptable toxicity. The initial cohorts of patients are treated with one course of either MHC Class I-binding or MHC Class II-binding peptides. If these Class I or Class II binding peptides are safe individually, subsequent cohorts of patients with appropriate HLA type receive both types of peptides in combination.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer with evidence of progressive disease despite hormonal therapy (i.e., hormone-refractory prostate cancer)

  * Metastatic disease
  * Progressive disease defined by any of the following:

    * New bone lesion on bone scan
    * Progression of nodal or soft tissue as evidenced by standard radiographic methods, i.e., CT scan or MRI
    * A 50% increase in PSA level from the nadir PSA level confirmed twice and measured at least 2 weeks apart, with stable and measurable disease
* Castrate serum levels of testosterone < 50 ng/dL
* If patient was receiving anti-androgen therapy, in addition to luteinizing hormone-releasing hormone (LHRH) agonist therapy, the evidence of progressive disease should persist after a trial of anti-androgen withdrawal

  * Treatment with LHRH agonist to maintain androgen ablation must continue throughout this trial
* Baseline PSA ≥ 10 ng/mL
* All patients with androgen-independent prostate cancer and matched HLA typing are eligible for vaccination regardless of initial NY-ESO-1 expression status

  * Patients must be typed for HLA-DR4, DR13, DP4, or HLA-A2 haplotypes
* No active brain metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 10 mg/dL
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* SGPT ≤ 3 times upper limit of normal
* Serum creatinine ≤ 2 mg/dL
* Wiling to be followed at Baylor College of Medicine
* No serious intercurrent medical illness
* No history of primary or secondary immunodeficiency
* No active systemic infection
* No known hepatitis B surface antigen, hepatitis C, or HIV antibody positivity
* No history of cardiac arrhythmia or ischemic heart disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior immunotherapy (including anti-androgen therapy) and recovered
* More than 28 days since prior chemotherapy
* No concurrent immunosuppressive drugs such as systemic corticosteroids

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Tolerability
Toxicity

SECONDARY OUTCOMES:
Immunological response

CONTACTS AND LOCATIONS:
Overall Officials: Teresa G. Hayes, MD, PhD, Study Chair — Veterans Affairs Medical Center - Houston
Locations (1):
- Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Sonpavde G, Wang M, Peterson LE, Wang HY, Joe T, Mims MP, Kadmon D, Ittmann MM, Wheeler TM, Gee AP, Wang RF, Hayes TG. HLA-restricted NY-ESO-1 peptide immunotherapy for metastatic castration resistant prostate cancer. Invest New Drugs. 2014 Apr;32(2):235-242. doi: 10.1007/s10637-013-9960-9. Epub 2013 Apr 23. PMID 23609828